CLINICAL TRIAL: NCT06902987
Title: Efficacy and Safety of Upatinib in the Treatment of Active Anal Fistulas in Crohn's Disease: a Single-center, Single-arm Study
Brief Title: Efficacy and Safety of Upatinib in the Treatment of Active Anal Fistulas in Crohn's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024ZSLYEC-371
Record Dates: First submitted 2025-01-02; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Crohn's Diseases; Active Anal Fistula; Upadacitinib
MeSH Terms: interventions — upadacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The primary endpoint was the combined response rate at 12 weeks of treatment (Other): Combined response refers to clinical response plus imaging response. Clinical response was defined as 100% closure of the external orifice of the fistula and no fluid seepage from the patient's complaint or physician's acupressure. Imaging remission was defined as the absence of > 2cm pyo-filling fistula on perianal MRI and the absence of edema and active inflammation. Clinical response for the primary endpoint was judged by two experienced senior physicians and, if inconsistent, by a third clinician. The imaging was judged by two senior doctors in the independent third party diagnostic team, and if the judgment was inconsistent, the third team physician made the judgment
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Enrolled patients received oral upatinib treatment with a conventional induction dose of 45mg/d for 12 weeks, followed by a maintenance dose of 15m/d or 30mg/d

SUMMARY:
Anal fistula is the most common perianal lesion of Crohn's disease (CD), and the incidence of anal fistula in eastern CD population is significantly higher than that in Western population. The treatment of CD active anal fistula is difficult, which seriously affects the quality of life of patients and consumes a lot of medical resources. Injection of biological agents is the most commonly used method for the treatment of CD anal fistula, small molecule drugs can be taken orally, and the curative effect is more lasting. Upadacitinib was the first small molecule drug approved for CD treatment in China on June 30, 2023. At present, there is only one post-subgroup analysis of a global Phase 3 clinical study on Upatinib in the treatment of CD anal fistula, and the number of active anal fistula cases included is small, and the study objects are mostly western populations. This study intends to include CD patients with active anal fistula, and adopts the method of single-center single-arm study to explore the efficacy of Upatinib in the treatment of CD anal fistula, so as to provide more evidence-based medical evidence for the drug selection of CD anal fistula in China.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic non-specific inflammatory disease of the intestine, and anal fistula is the most common perianal lesion in CD. Active anal fistula refers to the infection of the fistula, which causes perianal pain, discharge, redness, swelling, and even fever in patients. Biologics are currently the most widely used drugs for treating CD anal fistula. Studies with fistula healing as the main endpoint of observation show that the clinical remission rate of fistula is about 50% at most. CD anal fistula is difficult to treat, has a high recurrence rate, seriously affects the quality of life of patients, and consumes a large amount of medical resources.

CD anal fistula is a special subtype of CD, and exploring CD anal fistula has very important clinical significance. The incidence of anal fistula in Asian CD patients is significantly higher than that in Western CD patients; the prognosis of CD patients with anal fistula is worse, and the risk of intestinal stenosis or perforation is 3 to 4 times higher than that of patients without anal fistula; approximately 10% of patients present with anal fistula as the first manifestation of CD, and the symptoms of anal fistula most affect the quality of life of patients during the course of the disease; the susceptibility genes of CD anal fistula patients are different from those of other CD patients, and the susceptibility genes of the Asian CD population are different from those of the Western population. Our previous study included Han CD patients from southern China for analysis and found that polymorphisms in the IRGM, AOX1, and NKX2-3 genes are associated with the development of anal fistula.Compared with the widely used biologics for treating CD, small molecule drugs have great prospects. Biologics are complex proteins that require injection for treatment, have immunogenicity, are prone to secondary failure, and are relatively expensive. In contrast, small molecule drugs have a relatively small molecular weight, are easier to pass through cell membranes; have a short half-life and can be taken orally; have no antigenicity or immunogenicity, and have better sustained efficacy; and have lower production costs.

Upadacitinib was approved for the treatment of CD on June 30, 2023, and it is the first small molecule drug approved for CD treatment in China. The New England Journal of Medicine recently published the results of a phase 3 clinical study of upadacitinib for CD [8]: In the induction period study, the clinical remission rate of the upadacitinib 45 mg treatment group was higher than that of the placebo group (U-EXCEL study, 49.5% vs. 29.1%; U-EXCEED study, 38.9% vs. 21.1%), and the endoscopic response rate was also higher than that of the placebo group (U-EXCEL study, 45.5% vs. 13.1%; U-EXCEED study, 34.6% vs. 3.5%); in the maintenance period study (U-ENDURE), the clinical remission rates (37.3% and 47.6%) and endoscopic response rates (27.6% and 40.1%) of the upadacitinib 15 mg and 30 mg treatment groups at week 52 were both higher than those of the placebo group (15.1% and 7.3%). The above study results show that upadacitinib is effective in treating CD.However, as a new small molecule drug, the efficacy of upadacitinib for the special subtype of CD anal fistula is not clear.

JAK/STAT is involved in innate and adaptive immunity. After activation, the signal is rapidly transmitted from the membrane to the nucleus, and then cytokines are activated, white blood cell transport is promoted, and cell proliferation is initiated, triggering intestinal inflammation and playing an important role in the pathogenesis of CD. The JAK/STAT signaling pathway may also be an important pathogenic mechanism of CD anal fistula. Manreet et al. found that CD anal fistula patients have gene variations in the JAK/STAT signaling pathway [9]. Upadacitinib targets and inhibits JAK1. Mechanistically, it may be effective for CD anal fistula. At present, only post hoc subgroup analysis data from the aforementioned three clinical studies on CD (not yet published) are available. In these studies, the complete remission rates of patients with active fistulas treated with different doses of upadacitinib at week 52 were 25% (3/12) and 10% (1/10), respectively, which were superior to the placebo group (0%, 0/23 and 0/7). However, the number of active fistula cases included in this post hoc subgroup analysis was relatively small, and the study subjects were mostly Western populations. Therefore, more efficacy data on this new small molecule drug for CD fistulas in the Chinese population are needed.

Therefore, this study intends to include CD patients with active fistulas and use a single-arm clinical study approach to explore the efficacy of upadacitinib in treating Chinese CD fistula patients. This will prepare for subsequent randomized controlled trials (RCTs) to further investigate the efficacy of different doses of upadacitinib in treating fistulas and compare the efficacy of upadacitinib with other biological agents in treating fistulas, and also provide more evidence-based medical evidence for the drug selection of CD fistulas.

Our hospital is one of the largest inflammatory bowel disease centers in the country. Additionally, due to the reputation of the anorectal surgery department, it has gathered a large number of fistula patients, providing a guarantee for the number of cases in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤70 years;
* Make a clear diagnosis of CD according to the "Consensus Opinions on the Diagnosis and Treatment of Inflammatory Bowel Disease (Beijing, 2018)";
* The disease severity of CD was moderate and severe according to Crohn's diseaseactivityindex (CDAI), that is, CDAI score > 220.
* Complicated with active anal fistula, that is, on the basis of perianal MRI confirmation of anal fistula, the patient has perianal pain, fluid seepage and other symptoms, and the transanal surgeon judges that the symptoms are related to anal fistula activity;
* Patients with previous thrombosis, including deep vein thrombosis, pulmonary thromboembolism, atrial thrombosis, peripheral artery thrombosis and cerebral thrombosis confirmed by imaging;
* Informed consent. The subjects gave barrier-free informed consent, voluntarily participated in the clinical study and signed the informed consent.

Exclusion Criteria:

* History of allergy to the active ingredient of upatinib;
* Severe damage of liver and kidney function; Hemoglobin < 8g/L;
* History of malignant tumor;
* Patients with previous thrombosis;
* Neutrophil count < 1×109/L; , or lymphocyte count < 500×109/L;
* Patients with intestinal complications (including intestinal stricture with proximal intestinal dilation or intestinal fistula). Diagnosis based on CTE/MRE.
* Presence of enterostomy;
* With active severe infection (such as sepsis) or opportunistic infection (such as active tuberculosis, shingles);
* Pregnant or planning pregnancy.
* Patients with vaginal fistula;
* Patients with anorectal stenosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical response at 12 weeks of treatment | 12 weeks
  Clinical response was defined as 100% closure of the external orifice of the fistula and no fluid seepage from the patient's complaint or physician's acupressure
Imaging remission at 12 weeks of treatment | 12 weeks
  Imaging remission was defined as the absence of > 2 cm pyo-filling fistula on perianal MRI and the absence of edema and active inflammation

SECONDARY OUTCOMES:
The clinical response rate of anal fistula at week 12/48 of treatment. | 12 weeks、48 weeks
  Clinical response: At least 50% of the external openings with exudate upon digital pressure at baseline are closed
The clinical remission rate of anal fistula at week 12/48 of treatment. | 12 weeks、48 weeks
  Clinical remission: The patient has no symptoms of perianal fistula exudate, and 100% of the external openings show no exudate upon digital pressure by the doctor.
The imaging remission rate of anal fistula at week 12/48 of treatment | 12 weeks、48 weeks
  Imaging remission: No abscess fistula larger than 2 cm is found on perianal MRI, and there is no edema or active inflammation (judged blindly by one radiologist).
The Perianal Disease Activity Index score at week 12/48 of treatment | 12 weeks、48 weeks
  Perianal Disease Activity Index(PDAI) is the core tool for evaluating perianal lesions in Crohn's disease, with a total score ranging from 0 to 20. A higher score indicates more severe perianal disease activity and a poorer prognosis
The van Assche Magnetic Resonance Imaging (MRI) Score of anal fistula at week 12/48 of treatment. | 12 weeks、48 weeks
  van Assche Magnetic Resonance Imaging (MRI) Score is an imaging assessment tool for Crohn's disease intestinal lesions, with a total score of 0-30 points. High scores reflect more severe intestinal damage and poorer clinical outcomes.
The CAF-QoL score of anal fistula at week 12/48 of treatment. | 12 weeks、48 weeks
  Complex Anal Fistula Quality of Life Questionnaire of anal fistula is a specific assessment tool used to evaluate the quality of life in patients with anal fistula, with scores typically ranging from 0 to 60 points. Higher scores indicate greater impairment in quality of life and poorer clinical outcomes
The CDAI of CD at week 12/48 of treatment. | 12 weeks、48 weeks
  Crohn's Disease Activity Index(CDAI) is a tool for assessing the activity level of Crohn's disease, with a score range of 0 to 600. A higher score indicates a worse disease state.
The mucosal healing rate (SES-CD) at week 12/48 of treatment. | 12 weeks、48 weeks
  Simple Endoscopic Score for Crohn's Disease(SES-CD) is the core assessment tool for evaluating the severity of endoscopic lesions in Crohn's disease, with a total score ranging from 0 to 60 points. Higher scores directly reflect more severe mucosal damage and poorer clinical outcomes.
Safety evaluation within 56 weeks of treatment. | 56 weeks
  Safety was evaluated at each follow-up, with adverse events recorded. The safety assessments included the name, frequency, and severity of adverse events, vital signs, physical examination findings, and laboratory test results.

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth afflicated of Sun-yat sen university, Guangzhou, Guangdong, China